CLINICAL TRIAL: NCT01422005
Title: Simultaneous Bimanual Training to Improve Motor Function Post-Stroke
Brief Title: Study of the Recovery of Muscle Function in the Arm/Hand After a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-00118; R#: 11-00118 (Other: Institutional Review Board - NYU School of Medicine)
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Hemiparesis
Keywords: Rehabilitation; Fingers; Grasp; Hand; Strength; Brain Infraction; Hand Function; Post Stroke; Neural mechanisms; Motor Control; Motor Function
MeSH Terms: conditions — Stroke; Paresis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Simultaneous Bimanual training: Patients who have had either an acute/subacute and a Chronic stroke will get training on the devices.
  Interventions: Other: Simultaneous Bimanual training
- Control Group (Active Comparator): Conventional Occupational Therapy: Patients who have had either an acute/subacute and Chronic Stroke with hemiperisis will get conventional therapy.
  Interventions: Other: Conventional Occupational Therapy

INTERVENTIONS:
Other: Simultaneous Bimanual training — Patients who have had a stroke and are in the Device group will undergo 12 weeks of training using the devices.
  Patients who have had a stroke and are in the Control group, will undergo 12 weeks of conventional therapy.
  Other Names: Device group; Control group
  Arms: Experimental group
Other: Conventional Occupational Therapy — Conventional Occupational Therapy will be given to patients in the control group.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
The purpose of this study is to examine if practicing joint movements using specially designed devices can help in the recovery of muscle function in the arm/hand after a stroke. Subjects may qualify for participation in this study because they had a stroke and have had difficulty using their affected arm/hand ever since.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term adult disability in the United States, and hemiparesis is the most common motor impairment that frequently leads to persistent deficits in hand function. The mechanisms of recovery of hand motor function after stroke are poorly understood, and the protocols used in clinical practice lack a solid scientific rationale. The long-term objective of this research is to understand the neural mechanisms underlying the recovery of voluntary motor functions in brain-injured patients in order to provide a more objective and scientific basis to rehabilitation protocols used in clinical practice.

These devices will be used to facilitate the training of either unimanual or bimanual movements that can be used both in the acute and chronic post-stroke period, even when there is little active movement in the affected upper extremity. The specially designed mechanical devices (BAT, PST and WIFIT), Psychophysical methods using an instrumented glove, and electromyographic recordings from upper extremity muscles to investigate the following specific aims in patients with post-stroke hemiparesis will lead to:

* greater extensor muscle activation and out of synergy movement compared with unimanual training facilitated by an external agent (e.g. another person).
* Bimanual training with the specially designed mechanical devices (BAT, PST and WIFIT) over 6 weeks will produce greater functional recovery in the affected upper extremity in patients with post-stroke hemiparesis, compared with conventional therapy.
* The gains in motor control and function will be greater in patients who begin bimanual training in the acute post-stroke phase (0-6) months, compared with those that begin in the chronic post-stroke phase (> 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow study instructions and likely to complete all required visits; ability to comply with the therapy protocol as assessed by the investigator; must be English speaking.
* Subjects must have had a unilateral stroke

Exclusion Criteria:

* Severe upper extremity spasticity suggested by an Ashworth score of >3 at any joint, or restriction of full passive range of motion.
* Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition such as psychotic illness or severe depression.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* History of surgery or other significant injury to either upper extremity causing mechanical limitations that preclude task performance.
* Previous neurological illness such as head trauma, prior stroke, epilepsy, or demyelinating disease.
* Complicating medical problems such as uncontrolled hypertension, diabetes with signs of polyneuropathy, severe renal, cardiac or pulmonary disease, or evidence of other concurrent neurologic or orthopedic conditions precluding the subject from complying with the study protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Measurement of hand function | Day 1
  The outcome measures using the devices will include:
  * hand function
  * range of motion
  * stiffness
  * extent of impairment on the affected side
  * temperature differences between the two sides of the body, and
  * skin sensitivity to pressure.
  Testing of independent finger movements and grasp-release during a functional task will be measured using an instrumented glove with concurrent electromyographic and 3-D Motion analysis of joint movements and muscle activity patterns.

SECONDARY OUTCOMES:
Measurement of Hand Function | Day 84
  The outcome measures using the devices will include:
  * hand function
  * range of motion
  * stiffness
  * extent of impairment on the affected side
  * temperature differences between the two sides of the body, and
  * skin sensitivity to pressure.
  Testing of independent finger movements and grasp-release during a functional task will be measured using an instrumented glove with concurrent electromyographic and 3-D Motion analysis of joint movements and muscle activity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: John R Rizzo, MD, Principal Investigator — New York Univeristy School of Medicine
Locations (1):
- New York Univeristy School of Medicine, New York, New York, United States